CLINICAL TRIAL: NCT03566368
Title: Incidence and Impact of Cardiac Dysfunction in Isolated Traumatic Brain Injury Patients Requiring Surgical Intervention
Brief Title: Cardiac Dysfunction in Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, S. Bharath, Senior Resident, National Institute of Mental Health and Neuro Sciences, India
Other Study IDs: III, 3.02 Neurosciences
Record Dates: First submitted 2018-04-19; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Trauma, Head; Cardiac Complication
Keywords: Cardiac Dysfunction; Traumatic Brain Injury
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic | interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Isolated Traumatic Brain Injury Patients requiring emergency surgical intervention.
  Interventions: Diagnostic Test: Electrocardiogram; Diagnostic Test: Transthoracic Echocardiogram; Diagnostic Test: Cardiac enzyme - Troponin I Levels

INTERVENTIONS:
Diagnostic Test: Electrocardiogram — a 12 lead surface electrocardiogram taken after connecting limb and chest electrodes
  Other Names: ECG
Diagnostic Test: Transthoracic Echocardiogram — Transthoracic echocardiogram performed to evaluate Cardiac function in parasternal - long and short axis, Apical - 4 chamber and 5 chamber views.
  Other Names: ECHO
Diagnostic Test: Cardiac enzyme - Troponin I Levels — Blood sample - venous collected to measure blood troponin - I levels.
  Other Names: TROP-I

SUMMARY:
Patients with Head Injury have been associated with varying degree of cardiac dysfunction resulting in adverse events during emergency surgery and during recover from head injury. This study intends to study the incidence and impact of cardiac dysfunction using electrocardiogram, transthoracic echocardiogram and cardiac enzyme levels in head injury patients during and following emergency surgery. Our results will facilitate better management, guide specific therapy and help in prognostication in this group of patients.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a major public health concern and a leading cause of traumatic death worldwide. It contributes to significant mortality, morbidity and economic costs. TBI along with secondary insults have been associated with worse neurologic and clinical outcomes. Post-TBI hypotension (systolic blood pressure <90 mmHg) has been directly linked to mortality. Cardiac dysfunction has been documented in TBI and implicated as a cause for hypotensive episode during TBI surgery. However in majority of the situations, the cause is often unknown, and the treatment is empiric.

Abnormal electrocardiographic (ECG) findings are associated with various neurologic hemorrhages which includes TBI, where both ischemic-like changes and a variety of repolarization abnormalities have been described. These changes are thought to be secondary to sympathetic over-activity and autonomic imbalance, and are associated with dysfunction documented by transthoracic echocardiography and cardiac enzyme elevations. Despite the frequency with which TBI affects the general population and the high prevalence of secondary end-organ dysfunction after TBI, its potential impact on cardiac function has received little attention outside of case reports, small case series & retrospective studies. In our study, we intend to evaluate the incidence and impact of cardiac dysfunction on neurological outcomes in TBI.

Methodology: The proposed study is prospective and observational. After obtaining informed consent, Adult traumatic brain injury patients posted for surgery are recruited. Preoperatively patient's demographic and clinical parameters are recorded.Patient management are according to insitutional practice in lines with Brain Trauma Foundation guidelines. ECG, transthoracic ECHO and blood levels for Troponin I are tested. Intraoperatively, patient's hemodynamics are monitored with EV1000- FLOTRAC sensor using a Radial arterial and central venous line conitnuously and important time points during surgery are noted. Intraoperative drugs, fluids and any events are noted. In the postoperative period, the same physiological parameters including ECG, ECHO and Trop I are recorded for 7 days starting from the day of surgery.

The result from this study will help us understand the nature and the severity of cardiac dysfunction in head injured Indian patients requiring surgery. This will help us in improving our current practices of perioperative management and minimize secondary insults during the patients hospital stay resulting in better neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated TBI requiring surgery
* Surgery performed within 48 hours after insult

Exclusion Criteria:

* Presence of extracranial injuries (such as but not limited to orthopedic/ chest/ cardiac/ abdominal/ pelvis)
* Penetrating craniocerebral injury
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of head injury requiring emergency intracranial surgery presenting to National Institute of Mental health and Neurosciences.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2015-12-05 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Left Ventricular Ejection Fraction < 50% and change following surgery | Preoperative, Postoperative day 1, Postoperative day 2, Postoperative day 3, Postoperative day 4, Postoperative day 5, Postoperative day 6, Postoperative day 7.
  On ECHO performed using Ultrasonography (M-Turbo; Sonosite, Bothwell, WA, USA) using phased array transducer with a scanning frequency between 5 and 1 MHz - Ejection fraction calculated using simpson's Biplane method in 4 chamber and 2 chamber apical view.
Incidence of Left ventricular regional wall motion abnormality and change following surgery | Preoperative, Postoperative day 1, Postoperative day 2, Postoperative day 3, Postoperative day 4, Postoperative day 5, Postoperative day 6, Postoperative day 7.
  On ECHO performed using Ultrasonography (M-Turbo; Sonosite, Bothwell, WA, USA) using phased array transducer with a scanning frequency between 5 and 1 MHz - Presence of regional wall motion abnormality assessed in Parasternal - long and short axis, Apical 4,2 and 5 chamber views.

SECONDARY OUTCOMES:
ECG abnormality - Tachycardia | Preoperative, Postoperative day 1, Postoperative day 2, Postoperative day 3, Postoperative day 4, Postoperative day 5, Postoperative day 6, Postoperative day 7.
  ECG - heart rate > 100 min
ECG abnormality - Bradycardia | Preoperative, Postoperative day 1, Postoperative day 2, Postoperative day 3, Postoperative day 4, Postoperative day 5, Postoperative day 6, Postoperative day 7.
  ECG - heart rate < 60/ min
ECG abnormaltiy - Prolonged PR interval | Preoperative, Postoperative day 1, Postoperative day 2, Postoperative day 3, Postoperative day 4, Postoperative day 5, Postoperative day 6, Postoperative day 7.
  ECG - Prolonged PR Interval >200 ms
ECG abnormality - Prolonged QRS duration | Preoperative, Postoperative day 1, Postoperative day 2, Postoperative day 3, Postoperative day 4, Postoperative day 5, Postoperative day 6, Postoperative day 7.
  ECG - Prolonged QRS duration >120 ms
ECG abnormality - ST-T changes | Preoperative, Postoperative day 1, Postoperative day 2, Postoperative day 3, Postoperative day 4, Postoperative day 5, Postoperative day 6, Postoperative day 7.
  ECG - ST segment elevation and depression ≥0.1 mV in limb leads and ≥0.2 mV in chest leads, inverted (negative) T wave in any lead apart from aVR and V1
ECG abnormality - Morphological End Repolarization abnormalities | Preoperative, Postoperative day 1, Postoperative day 2, Postoperative day 3, Postoperative day 4, Postoperative day 5, Postoperative day 6, Postoperative day 7.
  ECG - T-wave showing biphasic, 2-peaked or separated U wave ≥0.1 mV
Elevated Cardiac Enzyme Levels | Preoperative, Postoperative day 1, Postoperative day 2, Postoperative day 3, Postoperative day 4, Postoperative day 5, Postoperative day 6, Postoperative day 7.
  TROP I levels tested by i-STAT cTnI method on i-STAT device (Abbott Diagnostics, Abbott Park, IL) > 0.1 ng/mL.
Short Term neurological outcome | Preoperative, Postoperative day 1, Postoperative day 2, Postoperative day 3, Postoperative day 4, Postoperative day 5, Postoperative day 6, Postoperative day 7, At 1 month.
  Glasgow coma score (3-15) recorded at bedside.
Hemodynamic Parameter - Cardiac Index | Continuous Values at 1 Min interval throughout the intraoperative period.
  Cardiac Index values obtained from FloTrac transducer (FloTracTM, Edwards Lifesciences, Irvine, CA, USA) was used to connect the arterial line to the EV1000 clinical platform (Edwards Lifesciences, Irvine, CA, USA).
Hemodynamic Parameter - Stroke volume index | Continuous Values at 1 Min interval throughout the intraoperative period.
  Stroke volume index values obtained from FloTrac transducer (FloTracTM, Edwards Lifesciences, Irvine, CA, USA) was used to connect the arterial line to the EV1000 clinical platform (Edwards Lifesciences, Irvine, CA, USA).
Hemodynamic parameter - Heart Rate | Continuous Values at 1 Min interval throughout the intraoperative period.
  Heart rate values obtained from FloTrac transducer (FloTracTM, Edwards Lifesciences, Irvine, CA, USA) was used to connect the arterial line to the EV1000 clinical platform (Edwards Lifesciences, Irvine, CA, USA).
Hemodynamic parameter - Mean Arterial Pressure | Continuous Values at 1 Min interval throughout the intraoperative period.
  Mean Arterial Pressure values obtained from FloTrac transducer (FloTracTM, Edwards Lifesciences, Irvine, CA, USA) was used to connect the arterial line to the EV1000 clinical platform (Edwards Lifesciences, Irvine, CA, USA).
Hemodynamic parameter - Stroke Volume Variation | Continuous Values at 1 Min interval throughout the intraoperative period.
  Stroke Volume Variation values obtained from FloTrac transducer (FloTracTM, Edwards Lifesciences, Irvine, CA, USA) was used to connect the arterial line to the EV1000 clinical platform (Edwards Lifesciences, Irvine, CA, USA).
Hemodynamic parameter - Systemic Vascular Resistance Index | Continuous Values at 1 Min interval throughout the intraoperative period.
  Systemic Vascular Resistance Index values obtained from FloTrac transducer (FloTracTM, Edwards Lifesciences, Irvine, CA, USA) was used to connect the arterial line to the EV1000 clinical platform (Edwards Lifesciences, Irvine, CA, USA).
Long term neurological outcome | At 3 Months, At 6 months, At 1 year.
  Extended Glasgow Outcome score (1-8)
Hospital Stay | At 1 month
  Total number of days in hospital from admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bharath Srinivasaiah, MD, Principal Investigator — National Institute of Mental Health and Neuro Sciences, India
Locations (1):
- National Institute of Mental Health and Neurosciences, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prathep S, Sharma D, Hallman M, Joffe A, Krishnamoorthy V, Mackensen GB, Vavilala MS. Preliminary report on cardiac dysfunction after isolated traumatic brain injury. Crit Care Med. 2014 Jan;42(1):142-7. doi: 10.1097/CCM.0b013e318298a890. PMID 23963125